CLINICAL TRIAL: NCT06991062
Title: Bayesian Neurobehavioral Phenotyping: From Mechanism Identification to Personalized Neuromodulation Treatments. R61 PHASE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-1316; NCI-2025-03773 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2025-05-22; First posted 2025-05-25 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FP1 (cTBS) then F3 (iTBS) (Experimental): Participants will be recruit using on-line, social media, radio, and print advertisements.
  Interventions: Procedure: Repetitive Transcranial Magnetic Stimulation (rTMS)
- F3 (iTBS) then Fp1 (cTBS) (Experimental): Participants will be recruit using on-line, social media, radio, and print advertisements.
  Interventions: Procedure: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Procedure: Repetitive Transcranial Magnetic Stimulation (rTMS) — TMS is a non-invasive procedure in which a coil is placed over the scalp, and focused magnetic pulses are applied to parts of the brain through the coil.

SUMMARY:
The goal of this clinical research study is to learn more about whether individual differences in brain responses to emotional triggers impact rTMS (repetitive transcranial magnetic stimulation) responses in people who smoke.

DETAILED DESCRIPTION:
Primary Objectives:

1. Determine the extent to which neuroaffective individual differences moderate rTMS treatment effects. Our working hypothesis is that smokers characterized by the LPP+ profile will be more likely to reduce nicotine self-administration after inhibitory rTMS to the VMPFC than after excitatory rTMS to the DLPFC.
2. Determine the extent to which neurocognitive individual differences moderate rTMS treatment effects. Our working hypothesis is that smokers characterized by the θ+ profile will be more likely to reduce nicotine self-administration after excitatory rTMS to the DLPFC than after inhibitory rTMS to the VMPFC.

Exploratory Objectives:

Our long-term goal is to develop image-guided, personalized rTMS interventions. Carefully assessing the time required for each step in the protocol will allow us to identify opportunities to further optimize our procedures and reduce visit duration in our future studies.

We will measure:

1. The time required by the staff to conduct each ERP assessment.
2. The time between the end of the last rTMS session and the start of the second ERP assessment.

We will analyze each measure to obtain an accurate estimate of the duration of each step in the procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21 to 60 years
2. Report smoking on average, 5 or more cigarettes, little cigars and/or cigarillos per day, within the past 30 days preceding the screening visit.
3. Expired carbon monoxide (CO) ≥ 6ppm and/or test positive for cotinine using a urine cotinine test on day of study visit.
4. Able to follow verbal and written instructions in English and complete all aspects of the study.
5. Have an address and telephone number where they may be reached.
6. Subjects must report current stable residence. Stable residence is a domicile in which an individual can operate as if it were their own homestead and does not include shelters, halfway houses, treatment centers, or group homes.
7. Meet safety criteria for EEG.
8. Be willing to vape from an e-cigarette during specified tasks.
9. Meet safety criteria for rTMS. Note that if a participant is not eligible for rTMS but is eligible for EEG, they may complete the EEG portion of the study.
10. Willing and able to independently remove any metal from the neck and above for rTMS procedures (e.g., jewelry)
11. Provides written informed consent and agree to all assessments and study procedures.
12. Agrees to complete telehealth (live audio-video conference and/or phone) and in-person visits and to be contacted via text.

    Exclusion Criteria:
13. rTMS exposure for treatment or research purposes in the last 6 months.
14. History of seizure, epilepsy, syncope, fainting episode, or head trauma resulting in loss of consciousness.
15. Presence or history of neurological disorders (migraine, stroke, Alzheimer's Disease and other Dementias, Parkinson's Disease, Multiple Sclerosis, Traumatic Brain Injury (TBI), increased intracranial pressure).
16. History of brain surgery, implanted electronic device, metal in the head.
17. Cardiac pacemakers, neural stimulators, implantable defibrillator, implanted medication pumps or sensors, intracardiac lines, or acute, unstable cardiac disease, with intracranial implants (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes)
18. History of or currently under medical care for myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke, or transient ischemic attack.
19. Reports vision problems that are not treated.
20. Has a hairstyle not compatible with the EEG and unwilling to modify hairstyle (e.g., braids, ponytails, dreadlocks, non-removable hair extensions or wigs, etc.) to accommodate the EGG net that is required to be worn on the scalp during the experimental procedure.
21. Reports current diagnosis or history of type I diabetes.
22. Currently using insulin.
23. Have undergone bariatric surgery.
24. Currently being enrolled in a weight loss program.
25. Takes any prescription or over the counter medications or supplements to control weight and/or appetite.
26. Self-report a history of or current diagnosis of a mental health condition.
27. Reports insomnia (<4 hours sleep per night, in 3 or more nights per week in the last 3 months)
28. Reports <4 hours of sleep the day of the visit
29. Reports using marijuana on a daily basis.
30. Reports having used any other illicit drugs (other than marijuana) or prescription medications for non-medical reasons in the last 12 months.
31. Currently receiving treatment for substance use disorder (e.g., alcohol, opioids, cocaine, marijuana, or stimulants).
32. Females who report averaging more than 7 alcoholic drinks, or males who report averaging more than 14 alcoholic drinks in a single week in the last 30 days.
33. Current use of certain medications (last 3 months):

    Investigational drugs. Drugs of anti or pro-convulsive action. Medications with psychotropic effects (e.g., antidepressants, antipsychotics).

    Medications known to increase risk of seizure Smoking cessation medication (e.g., Zyban, Wellbutrin, Wellbutrin SR, Chantix). Nicotine replacement therapy with the intent to quit smoking (e.g., patches, gum, lozenge, pouches, etc).
34. Being pregnant or lactating
35. Self-reported noise-induced hearing loss or tinnitus.
36. Currently participating in any other research study.
37. Any otherwise not specified medical or psychiatric condition, illness, disorder, or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator and/or Study Physician.

37. Any otherwise not specified medical or psychiatric condition, illness, disorder, or concomitant medication that could compromise participant safety or treatment, as determined by the Principal Investigator and/or Study Physician.

38. Subjects considered by the investigator as unsuitable for the study for reasons not otherwise stated.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Versace, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org